CLINICAL TRIAL: NCT00964392
Title: NAVISTAR® THERMOCOOL® Catheter for the Radiofrequency Ablation of Drug Refractory Recurrent Symptomatic Paroxysmal Atrial Fibrillation - Post Approval Registry
Brief Title: NAVISTAR® THERMOCOOL® Catheter Post Approval Registry
Acronym: AF Registry
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMA #P030031/S014
Record Dates: First submitted 2009-08-20; First posted 2009-08-24 (Estimated); Results first posted 2017-04-26 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- More-Experienced Physicians (MEP) (Experimental): Physicians who perform greater than or equal to 50 atrial fibrillation ablation procedures per year.
  Interventions: Procedure: Atrial fibrillation ablation
- Less-Experienced Physicians (LEP) (Experimental): Physicians who perform less than 50 atrial fibrillation ablation procedures per year.
  Interventions: Procedure: Atrial fibrillation ablation

INTERVENTIONS:
Procedure: Atrial fibrillation ablation — Radiofrequency ablation

SUMMARY:
The purpose of this registry is to provide additional corroborative short-term safety and long-term safety data for the NAVISTAR THERMOCOOL and NAVISTAR EZ STEER THERMOCOOL catheters in the treatment of symptomatic Paroxysmal Atrial Fibrillation (PAF).

DETAILED DESCRIPTION:
This registry is a prospective, multi-center, non-randomized post approval evaluation comprised of two (2) registry arms with independent hypotheses. The registry arms are defined as; Arm 1) physicians who perform greater than or equal to 50 atrial fibrillation ablation procedures per year and Arm 2) physicians who perform less than 50 atrial fibrillation ablation procedures per year. Subjects with drug refractory recurrent symptomatic PAF will be considered for this post approval registry. This registry will be conducted at up to 40 centers in a minimum of 381 evaluable subjects. The devices are currently FDA approved for commercial distribution under PMA #P030031/S11.

ELIGIBILITY:
Inclusion Criteria:

Candidates for this registry must meet ALL of the following criteria:

* Patients with drug refractory recurrent symptomatic PAF who have had three (3) AF episodes in the six (6) months prior to enrollment and one AF episode documented within the one (1) year prior to enrollment. Documentation may include electrocardiogram (ECG), transtelephonic monitor (TTM), Holter monitor (HM), or telemetry strip.
* Failure of at least one AAD for AF (class I or III or AV nodal blocking agent such as beta blockers and calcium channel blockers) as evidenced by recurrent symptomatic PAF, or intolerable side effects.
* Age 18 years or older.
* Able and willing to comply with all pre-, post- and follow-up testing and requirements.
* Signed Patient Informed Consent Form.

Exclusion Criteria:

Candidates will be excluded from the registry if any of the following conditions apply:

* Atrial fibrillation secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause.
* AF episodes that last longer than 30 days and are terminated via cardioversion.
* CABG procedure within the last six (6) months.
* Awaiting cardiac transplantation or other cardiac surgery.
* Documented left atrial thrombus on imaging (i.e., TEE, ICE, CT, or MRA).
* History of a documented thromboembolic event within the past one (1) year.
* Diagnosed atrial myxoma.
* Significant congenital anomaly or medical problem that in the opinion of the investigator would preclude enrollment in this registry.
* Women who are pregnant (by history of menstrual period or pregnancy test if the history is considered unreliable).
* Acute illness or active systemic infection or sepsis.
* Unstable angina.
* Uncontrolled heart failure.
* Myocardial infarction within the previous two (2) months.
* History of blood clotting or bleeding abnormalities.
* Contraindication to anticoagulation (i.e. heparin or warfarin).
* Life expectancy less than 12 months.
* Enrollment in an investigational study evaluating another device or drug.
* Presence of intramural thrombus, tumor or other abnormality that precludes catheter introduction or manipulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 437 (Actual)
Dates: Start 2009-09-01 (Actual); Primary Completion 2013-09-01 (Actual); Study Completion 2018-01-05 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was enrolled on September 29, 2009. Subject enrollment was completed and closed on October 01, 2013 after reaching a total of 437 enrolled (381 evaluable) subjects. The study is still ongoing. This report covers data up to the data download of June 23, 2015.
Groups:
- More-Experienced Physicians (MEP): MEP are defined as those who have performed greater than 50 AF ablation cases per year.
- Less-Experienced Physicians (LEP): LEP are defined as those who have performed less than or equal to 50 AF ablations per year.
Period: Overall Study
Arm/Group | More-Experienced Physicians (MEP) | Less-Experienced Physicians (LEP)
Started | 125 (Both safety and efficacy cohort: Total 128 (3 MEP Excluded)) | 282 (Both safety and efficacy cohort: Total 292 (10 LEP Excluded))
Completed | 72 | 92
Not Completed | 53 | 190
Not completed — Withdrawal by Subject | 4 | 6
Not completed — Lost to Follow-up | 4 | 10
Not completed — Early Termination, non-study arrhythmia | 1 | 6
Not completed — Not completed | 44 | 168

BASELINE CHARACTERISTICS:
Population: Enrolled subjects who have been assigned to MEP/LEP groups
Groups:
- More-experienced Physicians: Subjects were enrolled into sites where the primary investigators were more-experienced physicians (MEP). Those physicians were prospectively classified into the MEP group if he or she had performed greater than 50 atrial fibrillation (AF) ablation procedures per year.
- Less-experienced Physicians: Subjects were enrolled into sites where the primary investigators were less-experienced physicians (LEP). Those physicians were prospectively classified into the LEP group if he or she had performed less than or equal to 50 atrial fibrillation (AF) ablation procedures per year.
- Total: Total of all reporting groups
Arm/Group | More-experienced Physicians | Less-experienced Physicians | Total
Number analyzed (Participants) | 128 | 292 | 420
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (9.6) | 60.3 (9.5) | 60.5 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 102 | 146
  Male | 84 | 190 | 274
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 7 | 9
  Not Hispanic or Latino | 126 | 284 | 410
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 20 | 21
  White | 125 | 262 | 387
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 6 | 7
Region of Enrollment [Number; unit: participants]
  United States | 128 | 292 | 420

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Subjects Experiencing Primary Adverse Events Within Seven Days of the Ablation Procedure.
Description: The primary adverse events (AE) include Death, Myocardial infarction (MI), Pulmonary vein (PV) stenosis, Diaphragmatic paralysis, Atrio-esophageal fistula, Transient ischemic attack (TIA), Stroke/Cerebrovascular accident (CVA), Thromboembolism, Pericarditis, Cardiac tamponade, Pericardial effusion, Pneumothorax, Atrial perforation, Vascular access complications, Pulmonary edema, Hospitalization (including initial and prolonged, excluding those hospitalizations solely due to pre-existing arrhythmia recurrence), Heart block. Pulmonary vein stenosis (defined as ≥70% diameter reduction) and atrio-esophageal fistula occurring more than 7 days post-procedure shall be deemed a Primary AE. The primary endpoint for the Post-Approval Registry is a comparison of the 7-day primary AE rate against a performance criterion of 16 %. The 16% performance criterion is based on literature data and discussion with the FDA per IDE G030236.
Time Frame: Seven days post ablation procedure
Population: Safety population, which is defined as those subjects who underwent study catheter insertion. However subject LUC-030, who experienced one primary AE, was excluded from this analysis since the subject discontinued prior to RF ablation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | More-experienced Physicians | Less-experienced Physicians
Number analyzed (Participants) | 125 | 282
percentage of participants | 3.2 [0 to 7.2] | 6.4 [0 to 9.3]

2. Secondary Outcome: Percentage of Subjects Experienced Serious Adverse Events.
Description: The occurrence of serious adverse events (SAE) was used to provide the prospective long-term safety data. The SAEs are summarized by the following time periods: 0 to 30 days post-ablation, 31 days to 365 post-ablation, 366 to 730 days post-ablation, and more than 730 days post-ablation. One subject might have experienced SAEs in more than one time periods. This report covers the SAEs occurred from September 29, 2009 (first patient enrolled) to June 23, 2015 (data download date for this report).
Time Frame: First study day to 5 year post-ablation
Population: Safety population, which is defined as those subjects who underwent study catheter insertion. However subject LUC-030, who experienced one SAE, was excluded from this analysis since the subject discontinued prior to RF ablation.
Measure: Number; unit: percentage of participants
Arm/Group | More-experienced Physicians | Less-experienced Physicians
Number analyzed (Participants) | 125 | 282
percentage of participants
  1 to 30 days post-ablation | 6.4 | 12.1
  31 days to 365 days post-ablation | 11.2 | 14.5
  366 to 730 days post-ablation | 14.9 | 7.4
  More than 730 days post-ablation | 11.0 | 11.1

ADVERSE EVENTS:
Time Frame: Five years post-ablation
Arm/Group | More-experienced Physicians | Less-experienced Physicians
Serious Adverse Events (participants affected / at risk) | 41/125 | 95/282
Other Adverse Events (participants affected / at risk) | 78/125 | 168/282
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | More-experienced Physicians (N=125) | Less-experienced Physicians (N=282)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 7 (7)
Atrial flutter (Cardiac disorders) | 5 (7) | 4 (4)
Pericardial effusion (Cardiac disorders) | 2 (2) | 6 (6)
Chest pain (Cardiac disorders) | 4 (6) | 3 (3)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 3 (8)
Bradycardia (Cardiac disorders) | 4 (4) | 0 (0)
Syncope (Cardiac disorders) | 1 (1) | 3 (3)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 3 (3)
Dyspnoea (Cardiac disorders) | 2 (2) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 2 (2)
Fluid overload (Cardiac disorders) | 0 (0) | 2 (2)
Sick sinus syndrome (Cardiac disorders) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Arteriospasm coronary (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac perforation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac procedure complication (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Dizziness (Cardiac disorders) | 0 (0) | 1 (1)
Dressler's syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Presyncope (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Basedow's disease (Endocrine disorders) | 0 (0) | 1 (1)
Gastrinoma (Endocrine disorders) | 0 (0) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal injury (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia, obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Alcohol withdrawal syndrome (General disorders) | 0 (0) | 1 (1)
Device dislocation (General disorders) | 1 (2) | 0 (0)
Device related infection (General disorders) | 0 (0) | 1 (1)
Injection site haematoma (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Vessel puncture site haematoma (General disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 4 (5)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Biopsy thyroid gland abnormal (Investigations) | 1 (1) | 0 (0)
Cardiac pacemaker evaluation (Investigations) | 0 (0) | 1 (1)
Cardiac stress test abnormal (Investigations) | 1 (1) | 0 (0)
Heart rate increased (Investigations) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1)
Smear cervix abnormal (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain mass (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Myoclonus (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary vein stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 3 (3) | 3 (4)
Cardiac ablation (Surgical and medical procedures) | 0 (0) | 3 (3)
Cardiac pacemaker insertion (Surgical and medical procedures) | 1 (1) | 2 (2)
Hip arthroplasty (Surgical and medical procedures) | 1 (1) | 1 (1)
Abdominoplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Cancer surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Colectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Cryotherapy (Surgical and medical procedures) | 0 (0) | 1 (1)
Debridement (Surgical and medical procedures) | 0 (0) | 1 (1)
Implantable defibrillator replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
Knee operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Obesity surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Packed red blood cell transfusion (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 4 (4)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Artery dissection (Vascular disorders) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | More-experienced Physicians (N=125) | Less-experienced Physicians (N=282)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Ecchymosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 28 (44) | 44 (60)
Atrial flutter (Cardiac disorders) | 4 (4) | 14 (20)
Chest pain (Cardiac disorders) | 4 (5) | 13 (16)
Atrial tachycardia (Cardiac disorders) | 3 (3) | 8 (9)
Palpitations (Cardiac disorders) | 3 (3) | 7 (8)
Pericardial effusion (Cardiac disorders) | 3 (3) | 6 (6)
Dyspnoea (Cardiac disorders) | 4 (5) | 4 (4)
Chest discomfort (Cardiac disorders) | 3 (3) | 3 (3)
Dizziness (Cardiac disorders) | 1 (1) | 4 (4)
Arrhythmia (Cardiac disorders) | 2 (2) | 2 (2)
Oedema peripheral (Cardiac disorders) | 2 (2) | 2 (2)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 2 (2)
Dyspnoea exertional (Cardiac disorders) | 1 (1) | 2 (2)
Syncope (Cardiac disorders) | 2 (2) | 1 (1)
Fluid overload (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac flutter (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac procedure complication (Cardiac disorders) | 0 (0) | 1 (1)
Hypertrophic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Cardiac disorders) | 0 (0) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Basedow's disease (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Thyroid neoplasm (Endocrine disorders) | 1 (1) | 0 (0)
Thyroiditis (Endocrine disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 4 (4)
Ocular hyperaemia (Eye disorders) | 2 (2) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Periorbital haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Scleral haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Gastrointestinal disorders) | 0 (0) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 3 (3)
Erosive oesophagitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Procedural nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fungal oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gastroenteritis viral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lip disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatic carcinoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Procedural vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tongue biting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vessel puncture site haematoma (General disorders) | 3 (3) | 4 (4)
Procedural pain (General disorders) | 0 (0) | 3 (3)
Fatigue (General disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 2 (2)
Vessel puncture site haemorrhage (General disorders) | 1 (1) | 1 (1)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1)
Device malfunction (General disorders) | 1 (1) | 0 (0)
Device power source issue (General disorders) | 0 (0) | 1 (1)
Drug intolerance (General disorders) | 0 (0) | 1 (1)
Flank pain (General disorders) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 0 (0) | 1 (1)
Injection site haemorrhage (General disorders) | 1 (1) | 0 (0)
Mass (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0)
Swelling (General disorders) | 1 (1) | 0 (0)
Wound secretion (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis infective (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 6 (8)
Herpes zoster (Infections and infestations) | 2 (3) | 3 (3)
Sinusitis (Infections and infestations) | 0 (0) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Procedural headache (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Animal scratch (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Confusion postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site erythema (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb crushing injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Median nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Nerve compression (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skeletal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 2 (2) | 2 (2)
Blood pressure abnormal (Investigations) | 0 (0) | 1 (1)
Blood pressure decreased (Investigations) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 1 (1)
Culture urine positive (Investigations) | 0 (0) | 1 (1)
Echocardiogram (Investigations) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1)
Electrocardiogram abnormal (Investigations) | 0 (0) | 1 (1)
Endoscopy upper gastrointestinal tract normal (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Prostatic specific antigen increased (Investigations) | 1 (1) | 0 (0)
Sinus rhythm (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 7 (7)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 7 (7)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cervicobrachial syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 3 (3)
Dysarthria (Nervous system disorders) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 2 (2)
Agitation (Nervous system disorders) | 1 (1) | 0 (0)
Dysphonia (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (Nervous system disorders) | 0 (0) | 1 (1)
Phrenic nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Acute psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 2 (2) | 7 (7)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Testicular swelling (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (7)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Pulmonary vein stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Cardiac ablation (Surgical and medical procedures) | 5 (5) | 7 (8)
Cardioversion (Surgical and medical procedures) | 2 (2) | 5 (6)
Cardiac pacemaker battery replacement (Surgical and medical procedures) | 1 (1) | 1 (1)
Cataract operation (Surgical and medical procedures) | 0 (0) | 2 (5)
Abdominal hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Cardiac pacemaker insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Carpal tunnel decompression (Surgical and medical procedures) | 1 (1) | 0 (0)
Endotracheal intubation (Surgical and medical procedures) | 0 (0) | 1 (1)
Haemorrhoid operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1)
High frequency ablation (Surgical and medical procedures) | 0 (0) | 1 (1)
Incisional drainage (Surgical and medical procedures) | 0 (0) | 1 (1)
Meniscus operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Peripheral artery angioplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Skin neoplasm excision (Surgical and medical procedures) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 4 (4) | 6 (6)
Arteriovenous fistula (Vascular disorders) | 2 (2) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between the Principal Investigator (PI)/Institution and the Sponsor (or its agents) that restricts the PI's rights to discuss, present or publish trial results after the trial is completed. Please contact Biosense Webster, Inc. for additional information.